CLINICAL TRIAL: NCT04606823
Title: Evaluation of Clinical Performance of Ponto Implantation Using a Minimally Invasive Surgical Technique - a Prospective Multicentre Study
Brief Title: Ponto Implantation Using a Minimally Invasive Surgical Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC108
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm (Other): In this single-arm study the patients will be undergoing a minimally invasive surgery after which they will re-visit the clinic at five occasions for follow-up visits (1-3 extra compared to routine clinical practice at the hospitals) and complete a quality of life-questinnaire three months after surgery.
  Interventions: Procedure: Minimally invasive surgery; Other: Glasgow Benefit Inventory (GBI); Other: Additional follow-up visits after surgery

INTERVENTIONS:
Procedure: Minimally invasive surgery — The subjects will be implanted with a bone anchored hearing system using a minimally invasive surgery.
Other: Glasgow Benefit Inventory (GBI) — A quality of life-questionnaire is to be completed by the subjects at one occasion.
Other: Additional follow-up visits after surgery — There are 1-3 additional follow-up visits after surgery (compared to the routine clinical practice of the surgeons/clinics).

SUMMARY:
This multi-centre study funded by Oticon Medical AB will be conducted at seven hospitals across Europe (UK, Sweden, Denmark and the Netherlands). In total, 50 adult patients with a hearing loss that are already planned for treatment with a percutaneous (through the skin) bone-anchored hearing system (BAHS) will be included in the study.

The purpose of the study is to investigate the rate of successful BAHS use after implantation of the Ponto implant system using a minimally invasive surgical technique.

DETAILED DESCRIPTION:
This multi-centre study funded by Oticon Medical AB will be conducted at seven hospitals across Europe (UK, Sweden, Denmark and the Netherlands). In total, 50 adult patients with a hearing loss that are already planned for treatment with a percutaneous (through the skin) bone-anchored hearing system (BAHS) will be included in the study.

The purpose of the study is to investigate the rate of successful BAHS use after implantation of the Ponto implant system using a minimally invasive surgical technique. The implant, coupled to a skin-penetrating abutment, is implanted in the bone behind the ear and is later loaded with a sound processor which transforms sound waves to sound vibrations that can be sent directly to the inner ear via the skull bone. The primary objective of this study is to investigate the proportion of implant/abutment complexes providing a reliable anchorage for a sound processor three months after implantation/surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patient indicated for surgical intervention with a bone anchored hearing system
* Signed informed consent
* Adequate bone quality to allow for a Ponto implant insertion, as judged by the investigator, and an expected bone thickness above 5 mm, where no complications during surgery are expected
* Skin thickness of 12 mm or less at the implant site

Exclusion Criteria:

* Patient undergoing re-implantation
* Patient who are unable or unwilling to follow investigational procedures/requirements, e.g. to complete quality of life scales
* Known condition or previous treatment that could jeopardize skin condition and wound healing over time as judged by the investigator (e.g. uncontrolled diabetes, previous radiotherapy in the area of interest)
* Known medical condition that contraindicate surgery as judged by the investigator
* Known and/or planned pregnancy at time of surgery
* Any other known condition that the investigator determines could interfere with compliance or investigation assessments
* Simultaneous participation in another clinical investigation with pharmaceutical and/or medical device which might cause interference with investigation participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry Powell, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (7):
- Aalborg University Hospital, Aalborg, Denmark
- Netherlands (2):
  - Univerisity Medical Center Groningen, Groningen
  - Radboud University Medical Center, Nijmegen
- Sahlgrenska University Hospital, Gothenburg, Sweden
- United Kingdom (3):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Guy's and St Thomas' NHS Foundation Trust, London

REFERENCES:
- [Derived] Teunissen EM, Aukema TW, Banga R, Eeg-Olofsson M, Hol MKS, Hougaard DD, Tysome JR, Johansson ML, Svensson S, Powell HRF. Evaluation of Clinical Performance of Ponto Implantation Using a Minimally Invasive Surgical Technique-A Prospective Multicenter Study. Otol Neurotol. 2024 Oct 1;45(9):1037-1044. doi: 10.1097/MAO.0000000000004315. Epub 2024 Aug 26. PMID 39186326

RESULTS

PARTICIPANT FLOW:
Groups:
- Single-arm: In this single-arm study the patients undergo a minimally invasive surgery to recieve a bone anchored hearing system. After implantation, the patients re-visit the clinic at five occasions for follow-up visits (1-3 extra compared to routine clinical practice at the hospitals) and complete a quality of life-questinnaire three months after surgery.
Period: Overall Study
Arm/Group | Single-arm
Started | 52 (Patients enrolled in the study)
Completed | 51 (Patients included in Intention-To-Treat (ITT) population at study completion)
Not Completed | 1
Not completed — Delayed surgery, withdrawn | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: Implants
Arm/Group | Single-arm
Number analyzed (Participants) | 51
Number analyzed (Implants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 46
  Asian | 2
  Hispanic | 1
  Other | 2
Region of Enrollment [Number; unit: participants]
  Sweden | 6
  Netherlands | 14
  Denmark | 6
  United Kingdom | 25
BMI [Mean (Standard Deviation); unit: kg/m2] | 27.0 (4.2)
Smoking [Count of Participants; unit: Participants]
  Current smoker | 8
  History of smoking | 21
  No smoking | 22
Hearing loss indication [Count of Participants; unit: Participants] — Duplicate hearing loss indications were reported for four participantients (e.g. for different ears).
  Participants
    Conductive hearing loss | 15
    Mixed hearing loss | 25
    Sensorineural hearing loss | 3
    Single sided deafness | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Implants With Reliable Anchorage for a Sound Processor
Description: The variables assessed to determine reliable anchorage in the study are implant survival and stability, skin reactions, skin overgrowth and pain preventing use of the sound processor. For a positive outcome of the primary endpoint (reliable anchorage), the implant should be in place and stable without any adverse skin reactions, skin overgrowth or pain preventing usage of the sound processor.
Time Frame: 3 months after implant surgery
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Single-arm
Number analyzed (Participants) | 51
Number analyzed (Implants) | 52
Implants | 49

2. Secondary Outcome: Number of Implants With Reliable Anchorage for a Sound Processor
Description: The variables assessed to determine reliable anchorage in the study are implant survival and stability, skin reactions, skin overgrowth and pain preventing use of the sound processor. For a positive outcome (reliable anchorage), the implant should be in place and stable without any adverse skin reactions, skin overgrowth or pain preventing usage of the sound processor.
Time Frame: 12 months after implant surgery
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Single-arm
Number analyzed (Participants) | 51
Number analyzed (Implants) | 52
Implants | 46

3. Secondary Outcome: Implant Survival
Description: Implant survival will be assessed by the investigator by means of a Yes/No question: Implant in place [Yes/No]
Time Frame: 12 months after implant surgery
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Single-arm
Number analyzed (Participants) | 51
Number analyzed (Implants) | 52
Implants | 48

4. Secondary Outcome: Implant Stability
Description: Clinical assessment of implant stability by the investigator by means of a Yes/No question: Implant stable [Yes/No]
Time Frame: 12 months after implant surgery
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Single-arm
Number analyzed (Participants) | 51
Number analyzed (Implants) | 52
Implants | 48

5. Secondary Outcome: Holgers Score Distribution
Description: Distribution of Holgers score ratings assigned by investigator across all study visits. The Holgers score is used to grade skin reactions around the skin-penetrating abutment on a scale from 0 to 4, where 0 indicates a reaction-free area whereas 4 indicates a severe infection often requiring removal of the implant.
  The results are presented based on Holgers score distribution across all study visits, as well as separate for each study visit and for unplanned visits.
Time Frame: 9 days, 5 weeks, 3-, 6-, and 12 months after implant surgery, and unplanned visits
Population: The analysis is based on number of implants (one participant had two implants). The total number of visits varies between different time points due to missed visits, and all available data is reported. Holgers scores were reported in a total of 22 unplanned visits.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Single-arm
Number analyzed (Participants) | 51
Number analyzed (Visits) | 265
Visits
  All study visits : Holgers 0 | 205
  All study visits : Holgers 1 | 53
  All study visits : Holgers 2 | 6
  All study visits : Holgers 3 | 1
  All study visits : Holgers 4 | 0
  9 days : Holgers 0 | 35
  9 days : Holgers 1 | 17
  9 days : Holgers 2 | 0
  9 days : Holgers 3 | 0
  9 days : Holgers 4 | 0
  5 weeks : Holgers 0 | 40
  5 weeks : Holgers 1 | 8
  5 weeks : Holgers 2 | 1
  5 weeks : Holgers 3 | 0
  5 weeks : Holgers 4 | 0
  3 months : Holgers 0 | 36
  3 months : Holgers 1 | 12
  3 months : Holgers 2 | 1
  3 months : Holgers 3 | 0
  3 months : Holgers 4 | 0
  6 months : Holgers 0 | 38
  6 months : Holgers 1 | 6
  6 months : Holgers 2 | 1
  6 months : Holgers 3 | 0
  6 months : Holgers 4 | 0
  12 months : Holgers 0 | 43
  12 months : Holgers 1 | 4
  12 months : Holgers 2 | 1
  12 months : Holgers 3 | 0
  12 months : Holgers 4 | 0
  Unplanned visits : Holgers 0 | 13
  Unplanned visits : Holgers 1 | 6
  Unplanned visits : Holgers 2 | 2
  Unplanned visits : Holgers 3 | 1
  Unplanned visits : Holgers 4 | 0

6. Secondary Outcome: Max Holgers Score
Description: Max Holgers score rating per patient across study visits. The Holgers score is used to grade skin reactions around the skin-penetrating abutment on a scale from 0 to 4, where 0 indicates a reaction-free area whereas 4 indicates a severe infection often requiring removal of the implant.
Time Frame: 12 months after implant surgery
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Single-arm
Number analyzed (Participants) | 51
Number analyzed (Implants) | 52
Implants
  Holgers 0 | 17
  Holgers 1 | 29
  Holgers 2 | 5
  Holgers 3 | 1
  Holgers 4 | 0

7. Secondary Outcome: Mild/Adverse Skin Reaction
Description: Mild/Adverse skin reaction per patient across study visits, where adverse skin reaction is defined as Holgers ≥ 2 on at least one follow-up visit. The Holgers score is used to grade skin reactions around the skin-penetrating abutment on a scale from 0 to 4, where 0 indicates a reaction-free area whereas 4 indicates a severe infection often requiring removal of the implant.
Time Frame: 12 months after implant surgery
Population: as for outcome 5
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Single-arm
Number analyzed (Participants) | 51
Number analyzed (Visits) | 265
Visits
  No or minor skin reaction (Holgers 0-1) | 258
  Adverse skin reaction (Holgers 2-4) | 7

8. Secondary Outcome: IPS (Inflammation, Pain, Skin Height) Scores
Description: Distribution of IPS scores assigned by investigator across all study visits. The IPS scale is used to assess soft tissue status including inflammation (I), pain (P), and skin height (S) for a skin-penetrating implant, with scores ranging from 0 to 4 for the I-scale, and from 0 to 2 for the P- and S-scales. The IPS score is presented as [Ix Px Sx] with x being the individual score for each parameter. A higher score reflects a more severe complication.
  The results are presented based on IPS score distribution across all study visits, as well as separate for each study visit and unplanned visits.
Time Frame: 9 days, 5 weeks, 3-, 6- and 12 months after implant surgery, and unplanned visits
Population: The analysis is based on number of implants (one participant had two implants). The total number of visits varies between different time points due to missed visits, and all available data is reported.
  IPS scores were reported in a total of 22 unplanned visits. For one unplanned visit, only I- and P-scores were reported.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Single-arm
Number analyzed (Participants) | 51
Number analyzed (Visits) | 265
Visits
  All study visits : I-score 0 | 195
  All study visits : I-score 1 | 55
  All study visits : I-score 2 | 13
  All study visits : I-score 3 | 2
  All study visits : I-score 4 | 0
  All study visits : P-score 0 | 209
  All study visits : P-score 1 | 38
  All study visits : P-score 2 | 18
  All study visits : S-score 0 | 243
  All study visits : S-score 1 | 21
  All study visits : S-score 2 | 0
  9 days : I-score 0 | 29
  9 days : I-score 1 | 18
  9 days : I-score 2 | 5
  9 days : I-score 3 | 0
  9 days : I-score 4 | 0
  9 days : P-score 0 | 31
  9 days : P-score 1 | 14
  9 days : P-score 2 | 7
  9 days : S-score 0 | 51
  9 days : S-score 1 | 1
  9 days : S-score 2 | 0
  5 weeks : I-score 0 | 39
  5 weeks : I-score 1 | 8
  5 weeks : I-score 2 | 1
  5 weeks : I-score 3 | 1
  5 weeks : I-score 4 | 0
  5 weeks : P-score 0 | 39
  5 weeks : P-score 1 | 10
  5 weeks : P-score 2 | 0
  5 weeks : S-score 0 | 45
  5 weeks : S-score 1 | 4
  5 weeks : S-score 2 | 0
  3 months : I-score 0 | 37
  3 months : I-score 1 | 10
  3 months : I-score 2 | 2
  3 months : I-score 3 | 0
  3 months : I-score 4 | 0
  3 months : P-score 0 | 38
  3 months : P-score 1 | 7
  3 months : P-score 2 | 4
  3 months : S-score 0 | 42
  3 months : S-score 1 | 7
  3 months : S-score 2 | 0
  6 months : I-score 0 | 37
  6 months : I-score 1 | 6
  6 months : I-score 2 | 1
  6 months : I-score 3 | 1
  6 months : I-score 4 | 0
  6 months : P-score 0 | 41
  6 months : P-score 1 | 1
  6 months : P-score 2 | 3
  6 months : S-score 0 | 41
  6 months : S-score 1 | 4
  6 months : S-score 2 | 0
  12 months : I-score 0 | 41
  12 months : I-score 1 | 5
  12 months : I-score 2 | 2
  12 months : I-score 3 | 0
  12 months : I-score 4 | 0
  12 months : P-score 0 | 40
  12 months : P-score 1 | 5
  12 months : P-score 2 | 3
  12 months : S-score 0 | 45
  12 months : S-score 1 | 3
  12 months : S-score 2 | 0
  Unplanned visits : I-score 0 | 12
  Unplanned visits : I-score 1 | 8
  Unplanned visits : I-score 2 | 2
  Unplanned visits : I-score 3 | 0
  Unplanned visits : I-score 4 | 0
  Unplanned visits : P-score 0 | 20
  Unplanned visits : P-score 1 | 1
  Unplanned visits : P-score 2 | 1
  Unplanned visits : S-score 0 | 19
  Unplanned visits : S-score 1 | 2
  Unplanned visits : S-score 2 | 0

9. Secondary Outcome: Wound Healing
Description: Investigator assessment of wound being completely healed by means of a Yes/No question.
  The results are presented for each study visit and for unplanned visits.
Time Frame: 9 days, 5 weeks and 3 months after implant surgery, and unplanned visits
Population: Wound healing status was reported in a total of 17 unplanned visits.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Single-arm
Number analyzed (Participants) | 51
Number analyzed (Visits) | 167
Visits
  9 days : Yes | 37
  9 days : No | 15
  5 weeks : Yes | 45
  5 weeks : No | 4
  3 months : Yes | 48
  3 months : No | 1
  Unplanned visits : Yes | 15
  Unplanned visits : No | 2

10. Secondary Outcome: Skin Overgrowth
Description: Skin overgrowth over implant/abutment complex judged by the investigator by means of a Yes/No question.
  The results are presented for each study visit and for unplanned visits.
Time Frame: 9 days, 5 weeks, 3-, 6-, and 12 months after implant surgery, and unplanned visits
Population: The analysis is based on number of implants (one participant had two implants). The total number of visits varies between different time points due to missed visits, and all available data is reported. Assessment of skin overgrowth was reported in a total of 22 unplanned visits.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Single-arm
Number analyzed (Participants) | 51
Number analyzed (Visits) | 265
Visits
  9 days : Yes | 0
  9 days : No | 52
  5 weeks : Yes | 0
  5 weeks : No | 49
  3 months : Yes | 0
  3 months : No | 49
  6 months : Yes | 0
  6 months : No | 45
  12 months : Yes | 0
  12 months : No | 48
  Unplanned visits : Yes | 1
  Unplanned visits : No | 21

11. Secondary Outcome: Post-operative Events Around Abutment
Description: Assessment of post-operative events by investigator into five different categories: None, Bleeding and/or hematoma, Hair in-growth, Skin dehiscence around abutment, and Other.
  The results are presented based on post-operative event distribution across all study visits, as well as separate for each study visit and unplanned visits.
Time Frame: 9 days, 5 weeks, 3-, 6-, and 12 months after implant surgery, and unplanned visits
Population: The analysis is based on number of implants (one participant had two implants). The total number of visits varies between different time points due to missed visits, and all available data is reported.
  For one visit, two post-operative events were reported for the same implant. Post-operative events were reported in a total of 25 unplanned visits.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Single-arm
Number analyzed (Participants) | 51
Number analyzed (Visits) | 269
Visits
  All study visits: None | 240
  All study visits : Bleeding and/or hematoma | 3
  All study visits : Hair in-growth | 1
  All study visits : Skin dehiscence around abutment | 18
  All study visits : Other | 7
  9 days : None | 39
  9 days : Bleeding and/or hematoma | 0
  9 days : Hair in-growth | 0
  9 days : Skin dehiscence around abutment | 13
  9 days : Other | 0
  5 weeks : None | 45
  5 weeks : Bleeding and/or hematoma | 1
  5 weeks : Hair in-growth | 0
  5 weeks : Skin dehiscence around abutment | 2
  5 weeks : Other | 2
  3 months : None | 44
  3 months : Bleeding and/or hematoma | 1
  3 months : Hair in-growth | 0
  3 months : Skin dehiscence around abutment | 1
  3 months : Other | 3
  6 months : None | 43
  6 months : Bleeding and/or hematoma | 0
  6 months : Hair in-growth | 0
  6 months : Skin dehiscence around abutment | 2
  6 months : Other | 0
  12 months : None | 47
  12 months : Bleeding and/or hematoma | 0
  12 months : Hair in-growth | 1
  12 months : Skin dehiscence around abutment | 0
  12 months : Other | 0
  Unplanned visits : None | 22
  Unplanned visits : Bleeding and/or hematoma | 1
  Unplanned visits : Hair in-growth | 0
  Unplanned visits : Skin dehiscence around abutment | 0
  Unplanned visits : Other | 2

12. Secondary Outcome: Patient-perceived Presence of Pain Around Abutment
Description: Assessment of presence of patient-perceived pain by means of a Yes/No question to the subject.
Time Frame: 9 days, 5 weeks, 3-, 6-, and 12 months after implant surgery, and unplanned visits
Population: The analysis is based on number of implants (one participant had two implants). The total number of visits varies between different time points due to missed visits, and all available data is reported.
  Assessment of pain was reported in a total of 23 unplanned visits.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Single-arm
Number analyzed (Participants) | 51
Number analyzed (Visits) | 266
Visits
  All study visits : No | 204
  All study visits : Yes | 62
  9 days : No | 31
  9 days : Yes | 21
  5 weeks : No | 39
  5 weeks : Yes | 10
  3 months : No | 36
  3 months : Yes | 13
  6 months : No | 41
  6 months : Yes | 4
  12 months : No | 38
  12 months : Yes | 10
  Unplanned visits : No | 19
  Unplanned visits : Yes | 4

13. Secondary Outcome: Patient-perceived Presence of Numbness Around Abutment
Description: Assessment of presence of patient-perceived numbness by means of a Yes/No question to the patient.
Time Frame: 9 days, 5 weeks, 3-, 6-, and 12 months after implant surgery, and unplanned visits
Population: The analysis is based on number of implants (one participant had two implants). The total number of visits varies between different time points due to missed visits, and all available data is reported.
  Assessment of numbness was reported in a total of 23 unplanned visits.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Single-arm
Number analyzed (Participants) | 51
Number analyzed (Visits) | 266
Visits
  All study visits : No numbness | 254
  All study visits : Presence of numbness | 12
  9 days : No numbness | 48
  9 days : Presence of numbness | 4
  5 weeks : No numbness | 46
  5 weeks : Presence of numbness | 3
  3 months : No numbness | 46
  3 months : Presence of numbness | 3
  6 months : No numbness | 44
  6 months : Presence of numbness | 1
  12 months : No numbness | 48
  12 months : Presence of numbness | 0
  Unplanned visits : No numbness | 22
  Unplanned visits : Presence of numbness | 1

14. Secondary Outcome: Duration of Surgery
Description: Length of surgery measured in minutes.
Time Frame: 3 months after implant surgery
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Implants
Arm/Group | Single-arm
Number analyzed (Participants) | 51
Number analyzed (Implants) | 52
minutes | 10.0 (5.5)

15. Secondary Outcome: Sound Processor Usage
Description: Average sound processor usage time.
Time Frame: 12 months after implant surgery
Population: Participants using the sound processor daily at 12 months after surgery
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Single-arm
Number analyzed (Participants) | 45
hours per day | 13.0 (3.3)

16. Secondary Outcome: Subjective Benefit After Surgery
Description: The Glasgow Benefit Inventory (GBI) is a validated, 18-item patient-reported questionnaire that assesses changes in health-related quality-of-life following otorhinolaryngological (ENT) interventions. The questionnaire evaluates the perceived benefit after a procedure and generates a Total Score and three subscale scores: General (12 items), Social Support (3 items), and Physical Health (3 items). Each score ranges from -100 to +100, where positive values indicate improvement, negative values indicate deterioration, and zero reflects no change. The Total Score is calculated as the mean of all item scores (not a sum of subscale scores), while each subscale score is calculated as the mean of the items belonging to that subscale.
Time Frame: 3 months after surgery
Population: Number of participants answering the GBI questionnaire at 3 months
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Single-arm
Number analyzed (Participants) | 46
Score
  Total score | 26.8 (18.0)
  General score | 37.7 (24.7)
  Social support score | 9.1 (19.5)
  Physical support score | 1.45 (24.3)

ADVERSE EVENTS:
Time Frame: 12 months
Description: An adverse event (AE) is defined as any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in subjects, users or other persons, in the context of a clinical investigation, whether or not related to the investigational medical device.
Arm/Group | Single-arm
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 1/51
Other Adverse Events (participants affected / at risk) | 16/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-arm (N=51)
Pain (abdomen, back) (Nervous system disorders) | 1 (2) — Hospitalisation because of abdominal- and backpain (pre-existing abdominal aneurysm)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-arm (N=51)
Pain (Nervous system disorders) | 6 (7) — Pain around implant/abutment area.
Infection (Infections and infestations) | 4 (5) — Infection around abutment area.
Bleeding (Blood and lymphatic system disorders) | 3 (3) — Bleeding around abutment.
Inflammation (Skin and subcutaneous tissue disorders) | 3 (3) — Inflammation around abutment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT04606823/Prot_SAP_000.pdf